CLINICAL TRIAL: NCT07046702
Title: 68Ga-MY6349 PET/CT in Solid Tumors and Compared With 18F-FDG PET/CT
Brief Title: 68Ga-MY6349 PET/CT in Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMYY-2024KY252
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Trop2; PET/CT
Keywords: Solid tumor; Trop2; PET/CT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 68Ga-MY6349 — Each subject receives a single intravenous injection of 68Ga-MY6349 and undergoes PET/CT imaging within the specified time.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-MY6349 PET/CT to detect the Trop-2 expression of tumor lesions in patients with solid tumors and to identify patients benefiting from Trop-2 PET/CT.

DETAILED DESCRIPTION:
As a new trophoblast cell-surface antigen 2 (Trop-2) targeting PET radiotracer, 68Ga-MY6349 is promising as an excellent imaging agent applicable to various cancers. In this research, subjects with various types of tumors underwent contemporaneous 68Ga-MY6349 and standard-of-care imaging (18F-FDG) either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of standard-of-care imaging and 68Ga-MY6349 PET/CT were recorded by visual interpretation. The diagnostic accuracy of 68Ga-MY6349 was calculated and compared to standard-of-care imaging.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or older)
* patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report)
* patients who had scheduled both standard-of-care imaging and 68Ga-MY6349 PET/CT scans
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee

Exclusion Criteria:

* patients with pregnancy
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Audult patients with solid tumor who had scheduled both standard-of-care imaging and 68Ga-MY6349 PET/CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of PET/CT imaging with 68Ga-MY6349 for the non-invasive assessment of Trop2 expression in various cancer types. | 1 week
  Tumor Trop2 expression analysis in a fresh biopsy sample will be correlated to 68Ga-MY6349 tumor uptake, evaluated by measuring standardized uptake value (SUV) on the 68Ga-MY6349 PET/CT.

SECONDARY OUTCOMES:
Description of 68Ga-MY6349 uptake by measuring standardized uptake value (SUV) in various types of tumors | 1 week
  Standardized uptake value (SUV) of 68Ga-MY6349 PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.

OTHER OUTCOMES:
To investigate the superiority of 68Ga-MY6349 PET/CT over 18F-FDG PET/CT in some tumors through comparative analysis. | 2 weeks
  The numbers of positive primary and metastatic lesions of standard-of-care imaging (18F-FDG PET/CT) and 68Ga-MY6349 PET/CT were recorded by visual interpretation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No